CLINICAL TRIAL: NCT01335685
Title: An Open-Label, Dose-Escalation, Phase 1/2 Study of the Oral Form of Ixazomib (MLN9708), a Next-Generation Proteasome Inhibitor, Administered in Combination With a Standard Care Regimen of Melphalan and Prednisone in Patients With Newly Diagnosed Multiple Myeloma Requiring Systemic Treatment
Brief Title: Study of Oral Ixazomib in Combination With Melphalan and Prednisone in Participants With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16006; 2010-023772-71 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-14 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm A: Ixazomib 3.0 mg (Experimental): Ixazomib 3.0 mg, capsules, orally, on Days 1, 4, 8, 11, 22, 25, 29, 32 plus melphalan 9 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle for up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 23 maintenance cycles; overall up to 32 cycles [34 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm A: Ixazomib 3.7 mg (Experimental): Ixazomib 3.7 mg, capsules, orally, on Days 1, 4, 8, 11, 22, 25, 29, 32 plus melphalan 9 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 10 maintenance cycles; overall up to 19 cycles [21 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm B: Ixazomib 3.0 mg (Experimental): Ixazomib 3.0 mg, capsules, orally, on Days 1, 8, 15 plus melphalan 6 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1-4 in 28-day cycle for up to 13 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 15 maintenance cycles; overall up to 27 cycles [25 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm B: Ixazomib 4.0 mg (Experimental): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15 cycle plus melphalan 6 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1-4 in 28-day cycle for up to 13 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 49 maintenance cycles; overall up to 61 cycles [58 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm B: Ixazomib 5.5 mg (Experimental): Ixazomib 5.5 mg, capsules, orally, on Days 1, 8, 15 plus melphalan 6 mg/m^2, tablets orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1-4 in 28-day cycle for up to 13 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 12 maintenance cycles; overall up to 24 cycles [24 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm C: Ixazomib 3.0 mg (Experimental): Ixazomib 3.0 mg, capsules, orally, on Days 1, 8, 15, 22, and 29 plus melphalan 9 mg/m^2, tablets orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 30 maintenance cycles; overall up to 39 cycles [40 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm C: Ixazomib 4.0 mg (Experimental): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15, 22, and 29 plus melphalan 9 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 12 maintenance cycles; overall up to 21 cycles [24 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone
- Arm D: Ixazomib 4.0 mg (Experimental): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 22, and 29 plus melphalan 9 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally, on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 28 maintenance cycles; overall up to 37 cycles [38 months]).
  Interventions: Drug: Ixazomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
Drug: Melphalan — Melphalan tablets
Drug: Prednisone — Prednisone tablets

SUMMARY:
The purpose of this phase 1/2, open-label study was to evaluate the effect of oral formulation of Ixazomib when added to standard melphalan and prednisone (MP) treatment. Both phases of the study included participants who had newly diagnosed multiple myeloma and were ineligible for high-dose therapy plus stem cell transplantation because of age (≥65 years of age) or coexisting conditions and for whom standard MP treatment was indicated.

DETAILED DESCRIPTION:
The drug tested in this study was called ixazomib (MLN9708). Ixazomib was tested to treat the people with newly diagnosed multiple myeloma requiring systemic treatment who were not eligible for stem cell transplantation. This study determined the safety, tolerability, efficacy, quality of life (QOL), and pharmacokinetics (PK)/pharmacodynamics (PD) of ixazomib.

The study enrolled 61 patients. The study was conducted in 2 parts: 1) phase 1 dose escalation and 2) phase 2 expansion at maximum tolerated dose. Participants were enrolled to receive:

* Ixazomib 3.0 mg, 3.7 mg, 4.0 mg, or 5.5. mg depending on the treatment assignment

This multicenter trial was conducted in the Unites states, Canada, United Kingdom, Spain and Czech Republic. The overall time to participate in this study is 5.5 years. Participants made multiple visits to the clinic and were followed up every 16 weeks after end of treatment until disease progression if stopped treatment before disease progression and then every 16 weeks up to start of next therapy or death whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Is indicated with standard melphalan prednisone (MP) treatment and is not a candidate for high-dose therapy plus stem cell transplantation (HDT-SCT) for 1 of the following reasons: the participant is 65 years of age or older OR the participant is less than 65 years of age but has significant comorbid condition(s) that are likely to have a negative impact on tolerability of HDT-SCT
* Is diagnosed with symptomatic multiple myeloma or asymptomatic myeloma with myeloma-related organ damage according to standard criteria
* Has measurable disease as specified in study protocol
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Has adequate hematologic, liver, and renal function

Exclusion Criteria

* Has peripheral neuropathy that is greater or equal to Grade 2
* Has major surgery or radiotherapy within 14 days before the first dose of study drug
* Has uncontrolled infection requiring systematic antibiotics
* Has diarrhea (> Grade 1)
* Has prior systemic therapy for multiple myeloma, including investigational drugs (prior treatment with corticosteroids or localized radiation therapy dose not disqualify the participantt)
* Has central nervous system involvement
* Has cardiac status as described in protocol
* Has known gastrointestinal condition or procedure that could interfere with swallowing or the oral absorption of tolerance of IXAZOMIB - Diagnosis of smoldering multiple myeloma, Waldenstrom's macroglobulinemia, POEMS syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome
* Has Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Is diagnosed or treated for another malignancy within 2 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease with the exception of nonmelanoma skin cancer or any completely resected carcinoma in situ
* Has serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-06-27 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (20):
- United States (2):
  - Lebanon, New Hampshire
  - Morgantown, West Virginia
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Québec
- Czechia (2):
  - Brno
  - Prague
- Spain (6):
  - Badalona
  - Barcelona
  - Donostia / San Sebastian
  - Madrid
  - Salamanca
  - Seville
- United Kingdom (7):
  - Bournemouth
  - Brighton
  - Cambridge
  - London
  - Nottingham
  - Oxford
  - Uxbridge

REFERENCES:
- [Derived] San-Miguel JF, Echeveste Gutierrez MA, Spicka I, Mateos MV, Song K, Craig MD, Blade J, Hajek R, Chen C, Di Bacco A, Estevam J, Gupta N, Byrne C, Lu V, van de Velde H, Lonial S. A phase I/II dose-escalation study investigating all-oral ixazomib-melphalan-prednisone induction followed by single-agent ixazomib maintenance in transplant-ineligible newly diagnosed multiple myeloma. Haematologica. 2018 Sep;103(9):1518-1526. doi: 10.3324/haematol.2017.185991. Epub 2018 Jun 28. PMID 29954932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in United States Canada, United Kingdom, Spain, and Czech Republic from 27 June 2011 to 29 December 2016.
Pre-assignment Details: Participants with a diagnosis of multiple myeloma (previously untreated) were enrolled to receive ixazomib orally at various doses in Phase 1. Only Arm B: Ixazomib 4.0 mg continued in Phase 2.
Period: Overall Study
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Started | 7 | 4 | 3 | 26 | 5 | 6 | 4 | 6
Completed | 4 | 3 | 1 | 15 | 5 | 1 | 2 | 3
Not Completed | 3 | 1 | 2 | 11 | 0 | 5 | 2 | 3
Not completed — Study Terminated by Sponsor | 2 | 1 | 1 | 10 | 0 | 4 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Groups:
- Arm A: Ixazomib 3.0 - 3.7 mg: Ixazomib 3.0 - 3.7 mg, capsules, orally, on Days 1, 4, 8, 11, 22, 25, 29, 32 plus melphalan 9 mg/m^2, tablets, orally, on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 23 maintenance cycles; overall up to 32 cycles).
- Arm B: Ixazomib 3.0 - 5.5 mg: Ixazomib 3.0 - 5.5 mg, capsules, orally, on Days 1, 8, 15 plus melphalan 6 mg/m^2, tablets, orally, on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally, on Days 1-4 for in 28-day cycle for up to 13 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 49 maintenance cycles; overall up to 61 cycles).
- Arm C: Ixazomib 3.0 - 4.0 mg: Ixazomib 3.0 - 4.0 mg, capsules, orally, on Days 1, 8, 15, 22, and 29 plus melphalan 9 mg/m^2, tablets, orally, on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally, on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 30 maintenance cycles; overall up to 39 cycles).
- Arm D: Ixazomib 4.0 mg: Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 22, and 29 plus melphalan 9 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles in maintenance phase (up to 28 maintenance cycles; overall up to 37 cycles).
- Total: Total of all reporting groups
Arm/Group | Arm A: Ixazomib 3.0 - 3.7 mg | Arm B: Ixazomib 3.0 - 5.5 mg | Arm C: Ixazomib 3.0 - 4.0 mg | Arm D: Ixazomib 4.0 mg | Total
Number analyzed (Participants) | 11 | 34 | 10 | 6 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (6.68) | 74.3 (4.79) | 76.3 (4.27) | 73.2 (9.66) | 74.5 (5.60)
Age, Customized [Count of Participants; unit: Participants]
  <75 | 6 | 19 | 2 | 4 | 31
  >=75 | 5 | 15 | 8 | 2 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 5 | 3 | 23
  Male | 8 | 22 | 5 | 3 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Missing | 2 | 3 | 0 | 0 | 5
  Not Hispanic or Latino | 9 | 31 | 10 | 6 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 10 | 32 | 9 | 6 | 57
  Other | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 6 | 2 | 0 | 8
  Czech Republic | 6 | 8 | 0 | 1 | 15
  Spain | 3 | 15 | 7 | 5 | 30
  United Kingdom | 1 | 2 | 1 | 0 | 4
  United States | 1 | 3 | 0 | 0 | 4
Height [Mean (Standard Deviation); unit: cm] — Population: Height data was only available for 11, 33, 9 and 6 participants in the Arms A, B, C and D respectively.
  cm
    number analyzed (Participants) | 11 | 33 | 9 | 6 | 59
    (all) | 162.24 (7.872) | 162.68 (12.087) | 164.50 (11.413) | 160.50 (16.897) | 162.65 (11.615)
Weight at Baseline [Mean (Standard Deviation); unit: kg] | 70.58 (9.389) | 73.43 (16.642) | 72.77 (20.532) | 66.97 (21.404) | 72.17 (16.509)
Body Surface Area at Baseline [Mean (Standard Deviation); unit: m^2] — Body Surface Area (m^2) = square root [height (cm) x weight (kg) / 3600]. Population: Body Surface Area data was only available for 11, 33, 9 and 6 participants in the Arms A, B, C and D respectively.
  m^2
    number analyzed (Participants) | 11 | 33 | 9 | 6 | 59
    (all) | 1.782 (0.1426) | 1.813 (0.2638) | 1.799 (0.3337) | 1.718 (0.3650) | 1.795 (0.2638)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Ixazomib (Phase 1)
Description: The RP2D is the maximum tolerated dose (MTD) or less. The MTD is defined as the dose range at which ≤ 1 of 6 evaluable participants experience dose limiting toxicities (DLT) within the first 28 days of treatment (end of Cycle 1).
Time Frame: Cycle 1, phase 1 (Up to 42 days)
Population: Dose Limiting Toxicity population included participants who received at least 80% of doses of MLN9708 and melphalan during Cycle 1 in Arms A or all doses of MLN9708 and melphalan during Cycle 1 in Arm B, C, D, or experience a DLT in Cycle 1 in the phase 1 dose escalation portion.
Measure: Number; unit: mg
Groups:
- Arm D: Ixazomib 4.0 mg: Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 22, and 29 plus melphalan 9 mg/m^2, tablets, orally on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally on Days 1 to 4 in 42-day cycle for up to 9 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 28 maintenance cycles; overall up to 37 cycles).
Arm/Group | Arm A: Ixazomib 3.0 - 3.7 mg | Arm B: Ixazomib 3.0 - 5.5 mg | Arm C: Ixazomib 3.0 - 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 11 | 34 | 10 | 6
mg | 3 | 4 | 3 | 4

2. Primary Outcome: Very Good Partial Response (VGPR) or Better Response Rate (Phase 2)
Description: VGPR or better response rate is defined as percentage of participants with a complete response (CR) and very good partial response (VGPR). Per International Myeloma Working Group Uniform Response Criteria (IMWG), CR: 1) Negative immunofixation on the serum and urine, 2) Disappearance of any soft tissue plasmacytomas and 3) < 5% plasma cells in bone marrow. VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hour.
Time Frame: Day 1 of every other cycle from Day 1 of Cycle 2 (each cycle of 28 days) until death (Up to 5.5 years)
Population: The response-evaluable population is defined as participants who received at least 5 of 8 MLN9708 doses in Arm A, at least 2 of 3 MLN9708 doses in Arm B, at least 4 of 5 MLN9708 doses in Arm C, or at least 3 of 4 MLN9708 doses in Arm D and had measurable disease at baseline and at least 1 post-baseline response assessment.
Measure: Number; unit: percentage of participants
Groups:
- Arm B: Ixazomib 4.0 mg (RP2D): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15 plus melphalan 6 mg/m^2, tablets, orally, on Days 1 to 4 and prednisone 60 mg/m^2, tablets, orally, on Days 1 to 4 in 28-day cycle for up to 13 cycles in induction phase followed by ixazomib at dose last tolerated in induction, orally, on Days 1, 8, 15 in 28-day cycle up to 12 cycles or until disease progression or unacceptable toxicity if deriving benefit in maintenance phase (up to 49 maintenance cycles; overall up to 61 cycles [58 months]).
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 23
percentage of participants | 48

3. Secondary Outcome: Maximum Inhibition Rate (Emax) (Phase 1)
Description: Whole blood 20S proteasome inhibition parameters
Time Frame: At multiple time points during Cycles 1-3 of each phase and arm of the study, throughout approximately 84-126 days depending on the arm of the study
Population: Due to the change in the planned analysis, the efficacy endpoint of maximum inhibition rate was not performed.
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time of Occurrence of Emax (TEmax) (Phase 1)
Description: Whole blood 20S proteasome inhibition parameters
Time Frame: as for outcome 3
Population: The efficacy endpoint of maximum inhibition rate was not performed due to the change in the planned analysis.
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib (Phase 1)
Time Frame: Pre-dose on Day 1 and at multiple timepoints (up to 8 hours) on Day 11 for Arm A, Day 15 for Arm B and Day 29 for Arms C and D
Population: The pharmacokinetics (PK) population consisted of all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of ixazomib PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 1 | 3 | 20 | 4 | 6 | 4 | 5
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 7 | 1 | 2 | 18 | 4 | 6 | 4 | 5
  Cycle 1, Day 1 | 26.791 (18.2608) | 39.300 (NA) — Standard deviation was not estimable for 1 participant. | 22.950 (NA) — Standard deviation was not estimable for 1 participant. | 53.278 (41.1963) | 104.225 (46.9148) | 55.367 (43.8052) | 50.875 (20.6487) | 72.080 (54.3984)
  Cycle 1, Day 11: number analyzed (Participants) | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11 | 69.214 (30.1985) | 22.000 (NA) — Standard deviation was not estimable for 1 participant. |  |  |  |  |  |
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 0 | 1 | 14 | 1 | 0 | 0 | 0
  Cycle 1, Day 15 |  |  | 30.267 (13.7173) | 85.636 (64.6346) | 285.000 (NA) — Standard deviation was not estimable for 1 participant. |  |  |
  Cycle 1, Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4
  Cycle 1, Day 29 |  |  |  |  |  | 59.560 (37.2229) | 109.000 (NA) — Standard deviation was not estimable for 2 participants. | 146.400 (90.1703)

6. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib (Phase 1)
Time Frame: as for outcome 5
Population: The PK population consisted of all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of ixazomib PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 1 | 3 | 20 | 4 | 6 | 4 | 5
hours
  Cycle 1, Day 1: number analyzed (Participants) | 7 | 1 | 2 | 18 | 4 | 6 | 4 | 5
  Cycle 1, Day 1 | 1.020 [0.617 to 4.000] | 0.517 [0.517 to 0.517] | 1.750 [1.470 to 2.030] | 1.000 [0.500 to 2.170] | 1.302 [0.533 to 4.000] | 1.560 [0.483 to 4.000] | 1.282 [0.500 to 4.000] | 0.567 [0.417 to 2.150]
  Cycle 1, Day 11: number analyzed (Participants) | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11 | 1.050 [0.500 to 4.000] | 8.000 [8.000 to 8.000] |  |  |  |  |  |
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 0 | 3 | 14 | 1 | 0 | 0 | 0
  Cycle 1, Day 15 |  |  | 0.833 [0.583 to 2.000] | 1.000 [0.500 to 4.000] | 0.500 [0.500 to 0.500] |  |  |
  Cycle 1, Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4
  Cycle 1, Day 29 |  |  |  |  |  | 1.500 [0.500 to 4.030] | 1.275 [0.550 to 2.000] | 0.760 [0.300 to 1.430]

7. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-time Curve Over the Dosing Interval for Ixazomib (Phase 1)
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 1 | 3 | 20 | 4 | 6 | 4 | 5
hr*ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 7 | 1 | 2 | 17 | 4 | 6 | 4 | 5
  Cycle 1, Day 1 | 319.714 (104.6721) | 287.000 (NA) — Standard deviation was not estimable for 1 participant. | 450.000 (NA) — Standard deviation was not estimable for 1 participant. | 806.824 (472.7173) | 1612.250 (1009.5816) | 662.833 (414.5178) | 1037.500 (397.8748) | 934.800 (390.2598)
  Cycle 1, Day 11: number analyzed (Participants) | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11 | 1227.143 (338.9550) | 1180.000 (NA) — Standard deviation was not estimable for 1 participant. |  |  |  |  |  |
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 0 | 3 | 14 | 1 | 0 | 0 | 0
  Cycle 1, Day 15 |  |  | 705.667 (92.5005) | 1610.500 (770.2156) | 1680.000 (NA) — Standard deviation was not estimable for 1 participant. |  |  |
  Cycle 1, Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4
  Cycle 1, Day 29 |  |  |  |  |  | 1527.800 (975.9914) | 2680.000 (NA) — Standard deviation was not estimable for 2 participants. | 2435.000 (1107.5047)

8. Secondary Outcome: Terminal Elimination Rate Constant (λz) for Ixazomib (Phase 1)
Description: Terminal elimination rate constant, calculated as the negative of the slope of the log-linear regression of the natural logarithm concentration-time curve during the terminal phase.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 1 | 3 | 20 | 4 | 6 | 4 | 5
1/hour
  Cycle 1, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0
  Cycle 1, Day 15 |  |  | 0.004 (NA) — Standard deviation was not estimable for 1 participant. | 0.006 (0.0018) | 0.007 (NA) — Standard deviation was not estimable for 3 participants. | NA (NA) — Standard deviation was not estimable for 1 participant. |  |
  Cycle 1, Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4
  Cycle 1, Day 29 |  |  |  |  |  | 0.005 (0.0021) | 0.005 (NA) — Standard deviation was not estimable for 2 participants. | 0.006 (0.0025)

9. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for Ixazomib (Phase 1)
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 1 | 3 | 20 | 4 | 6 | 4 | 5
hours
  Cycle 1, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0
  Cycle 1, Day 15 |  |  | 167.000 (NA) — Standard deviation was not estimable for 1 participant. | 130.362 (45.0672) | 98.900 (NA) — Standard deviation was not estimable for 3 participants. | NA (NA) — Standard deviation was not estimable for 1 participant. |  |
  Cycle 1, Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4
  Cycle 1, Day 29 |  |  |  |  |  | 140.575 (49.3760) | 163.500 (NA) — Standard deviation was not estimable for 2 participants. | 120.050 (45.6024)

10. Secondary Outcome: Observed Accumulation Ratio for AUCtau (Rac) (Phase 1)
Description: Accumulation ratio for AUCtau (Rac) was calculated as area under the curve from time zero to end of dosing interval (AUCtau) on Day 14 divided by area under the curve from time zero to end of dosing interval (AUCtau) on Day 1.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 1 | 3 | 20 | 4 | 6 | 4 | 5
ratio
  Cycle 1, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11: number analyzed (Participants) | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1, Day 11 | 4.019 (1.1349) | 4.120 (NA) — Standard deviation was not estimable for 1 participant. |  |  |  |  |  |
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 0 | 2 | 12 | 1 | 0 | 0 | 0
  Cycle 1, Day 15 |  |  | 1.700 (NA) — Standard deviation was not estimable for 2 participants. | 2.288 (0.6246) | 1.970 (NA) — Standard deviation was not estimable for 1 participant. |  |  |
  Cycle 1, Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4
  Cycle 1, Day 29 |  |  |  |  |  | 2.632 (0.6732) | 2.560 (NA) — Standard deviation was not estimable for 2 participants. | 2.540 (0.2061)

11. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with overall response including CR, VGPR, and partial response (PR). Per IMWG criteria, CR:1)Negative immunofixation on serum and urine, 2)Disappearance of any soft tissue plasmacytomas, 3)< 5% plasma cells in bone marrow. VGPR: Serum+urine M-protein detectable by immunofixation but not on electrophoresis/ 90% or >reduction in serum M-protein + urine M-protein level < 100 mg/ 24-hour. PR:1)≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24-hour. If serum+urine M-protein are unmeasurable, ≥50% decrease in difference between involved and uninvolved FLC levels is required. If serum+urine M-protein are unmeasurable and serum free light assay is also unmeasurable, ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was ≥30%. In addition, if present at baseline, a ≥50% reduction in size of soft tissue plasmacytomas is required.
Time Frame: Day 1 of every other cycle from Day 1 of Cycle 2 (each cycle of 28 days) up to 61 cycles, at end of treatment (Up to 5.5 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 3 | 3 | 23 | 5 | 5 | 3 | 4
percentage of participants | 86 [42 to 100] | 67 [9 to 99] | 100 [29 to 100] | 65 [43 to 84] | 60 [15 to 95] | 40 [5 to 85] | 67 [9 to 99] | 50 [7 to 93]

12. Secondary Outcome: Time to First Response (Phase 2)
Description: Response is defined as CR, VGPR and PR. Per IMWG criteria, CR:1)Negative immunofixation on serum+urine, 2)Disappearance of any soft tissue plasmacytomas, 3)< 5% plasma cells in bone marrow. VGPR: Serum+urine M-protein detectable by immunofixation but not on electrophoresis/ 90% or >reduction in serum M-protein + urine M-protein level < 100 mg/ 24-hour. PR:1)≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24-hour. If serum+urine M-protein are unmeasurable, ≥50% decrease in difference between involved and uninvolved FLC levels is required. Else, ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was ≥30%. In addition, if present at baseline, a ≥50% reduction in size of soft tissue plasmacytomas is required.
Time Frame: From the date of enrollment to the date of the first documented response for up to 5.5 years
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 15
months | 1.9 [1 to 7]

13. Secondary Outcome: Duration of Response (DOR) (Phase 2)
Description: DOR is defined as time of first documentation of a confirmed PR or better response to first documented PD or start of alternative therapy. DOR was presented for those achieving CR+VGPR+PR. Per IMWG criteria, CR:1)Negative immunofixation on serum+urine, 2)Disappearance of any soft tissue plasmacytomas, 3)< 5% plasma cells in bone marrow. VGPR: Serum+urine M-protein detectable by immunofixation but not on electrophoresis/ 90% or >reduction in serum M-protein + urine M-protein level < 100 mg/ 24-hour. PR:1)≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24-hour. If serum+urine M-protein are unmeasurable, ≥50% decrease in difference between involved and uninvolved FLC levels is required. Else, ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was ≥30%. In addition, if present at baseline, a ≥50% reduction in size of soft tissue plasmacytomas is required.
Time Frame: From the time from the date of first documentation of PR or better to the date of first documented disease progression for up to 5.5 years
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 23
months | 25.2 [4.6 to NA] — Lower limit of CI was not reached due to low number of participants with events.

14. Secondary Outcome: Time to Progression (TTP) (Phase 2)
Description: TTP is defined as time from date of enrollment to date of first documented disease progression (PD). Per IMWG criteria, progressive disease requires any 1 or more of following: Increase of ≥25% from nadir in serum M-component and/or (absolute increase must be ≥0.5 g/dL), urine M-component and/or (absolute increase must be ≥200 mg/24 hour. Participants without measurable serum+urine M-protein levels: difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dL. Bone marrow plasma cell percentage: absolute % must be ≥10%. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.85 mmol/L) that can be attributed solely to plasma cell proliferative disorder.
Time Frame: From the date of enrollment to the date of the first documented disease progression for up to 5.5 years
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 26
months | 22.1 [8.77 to NA] — Lower limit of CI was not reached due to low number of participants with events.

15. Secondary Outcome: Time to Next Therapy (Phase 2)
Description: Time to Next Therapy is defined as time from the date of enrollment to the date of subsequent antineoplastic therapy.
Time Frame: From the date of enrollment to the date of subsequent antineoplastic therapy for up to 5.5 years
Population: Time to next therapy was not analyzed due to the change in the planned analysis.
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 0

16. Secondary Outcome: Progression Free Survival (Phase 2)
Description: Progression Free Survival is defined as time in months from start of study treatment to first documentation of objective tumor progression per investigator assessment or up to death due to any cause, whichever occurs first. Per IMWG criteria, progressive disease requires any 1 or more of following: Increase of ≥25% from nadir in serum M-component and/or (absolute increase must be ≥0.5 g/dL), urine M-component and/or (absolute increase must be ≥200 mg/24 hour. Participants without measurable serum+urine M-protein levels: difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dL. Bone marrow plasma cell percentage: absolute % must be ≥10%. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.85 mmol/L) that can be attributed solely to plasma cell proliferative disorder.
Time Frame: From the date of enrollment to the date of the first documented disease progression or death due to any cause for up to 5.5 years
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 26
months | 18.4 [8.31 to 38.67]

17. Secondary Outcome: Overall Survival (Phase 2)
Description: Overall Survival is the time in months from start of study treatment to date of death due to any cause.
Time Frame: From date of enrollment to date of death, approximately 5.5 years (Approximate median follow-up: 43.6 months)
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 26
months | NA [34.99 to NA] — Median and lower limit of CI was not reached due to low number of participants with events.

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: From first dose of study drug through 30 days after last dose of study drug or until the start of subsequent antineoplastic therapy for up to 5.6 years
Population: The safety population consisted of participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Number analyzed (Participants) | 7 | 4 | 3 | 26 | 5 | 6 | 4 | 6
participants
  During Entire Study Any Adverse Event | 7 | 4 | 3 | 26 | 5 | 6 | 4 | 6
  Grade 3 or Higher Adverse Event | 7 | 4 | 3 | 21 | 5 | 5 | 4 | 5
  Serious Adverse Event | 2 | 4 | 3 | 12 | 3 | 4 | 2 | 1
  Adverse Event With Any Study Drug Discontinuation | 0 | 0 | 0 | 8 | 2 | 2 | 1 | 2
  Adverse Event With Any Study Drug Reduction | 4 | 2 | 1 | 13 | 3 | 3 | 2 | 4

19. Secondary Outcome: Assessments of Quality of Life (Phase 2)
Time Frame: Baseline, Day 1 of each treatment cycle, and Day 1 of each maintenance cycle, up to 5.5 years
Population: Assessments of quality of life parameters were not analyzed due to change in planned analysis.
Arm/Group | Arm B: Ixazomib 4.0 mg (RP2D)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after last dose of study drug or until the start of subsequent antineoplastic therapy for up to 5.6 years
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Arm A: Ixazomib 3.0 mg | Arm A: Ixazomib 3.7 mg | Arm B: Ixazomib 3.0 mg | Arm B: Ixazomib 4.0 mg | Arm B: Ixazomib 5.5 mg | Arm C: Ixazomib 3.0 mg | Arm C: Ixazomib 4.0 mg | Arm D: Ixazomib 4.0 mg
Serious Adverse Events (participants affected / at risk) | 2/7 | 4/4 | 3/3 | 12/26 | 3/5 | 4/6 | 2/4 | 1/6
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 3/3 | 26/26 | 5/5 | 6/6 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ixazomib 3.0 mg (N=7) | Arm A: Ixazomib 3.7 mg (N=4) | Arm B: Ixazomib 3.0 mg (N=3) | Arm B: Ixazomib 4.0 mg (N=26) | Arm B: Ixazomib 5.5 mg (N=5) | Arm C: Ixazomib 3.0 mg (N=6) | Arm C: Ixazomib 4.0 mg (N=4) | Arm D: Ixazomib 4.0 mg (N=6)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 — One treatment-emergent death occurred in Arm B during treatment with ixazombib 4.0 mg and is not related.
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred in Arm B during treatment with ixazombib 4.0 mg and is not related.
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred in Arm B during treatment with ixazombib 4.0 mg and is not related.
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ixazomib 3.0 mg (N=7) | Arm A: Ixazomib 3.7 mg (N=4) | Arm B: Ixazomib 3.0 mg (N=3) | Arm B: Ixazomib 4.0 mg (N=26) | Arm B: Ixazomib 5.5 mg (N=5) | Arm C: Ixazomib 3.0 mg (N=6) | Arm C: Ixazomib 4.0 mg (N=4) | Arm D: Ixazomib 4.0 mg (N=6)
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 1 | 17 | 5 | 2 | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 2 | 2 | 11 | 3 | 3 | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4 | 1 | 11 | 4 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 2 | 6 | 3 | 3 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 5 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue eruption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4 | 2 | 16 | 3 | 5 | 4 | 6
Neutropenia (Blood and lymphatic system disorders) | 5 | 4 | 2 | 12 | 2 | 2 | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 1 | 9 | 5 | 3 | 3 | 4
Lymphopenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 8 | 2 | 3 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 7 | 2 | 2 | 2 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 3 | 1 | 9 | 2 | 1 | 2 | 3
Pyrexia (General disorders) | 3 | 3 | 1 | 6 | 2 | 1 | 0 | 3
Fatigue (General disorders) | 6 | 0 | 1 | 9 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 7 | 2 | 2 | 3 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic fatigue syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 10 | 1 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 5 | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 6 | 0 | 3 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 6 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 4 | 2 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood electrolytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0 | 6 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 0 | 4 | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Peripheral coldness (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 9 | 0 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 2
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 1 | 8 | 3 | 0 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2 | 0 | 7 | 2 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 4 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 0 | 5 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 3 | 0 | 3 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 6 | 2 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 4 | 0 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property